CLINICAL TRIAL: NCT00944060
Title: A Pilot Study of Diabetes Risk Reduction Program With Overweight WIC Mothers
Brief Title: A Pilot Study of Diabetes Risk Reduction Program With WIC Mothers(The Special Supplemental Nutrition Program for Women, Infants, and Children) Overweight WIC Mothers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Purpose: Prevention
Other Study IDs: DK74511 (completed); 1R34DK074511-01A1 (NIH)
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Prevention of Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle intervention (Experimental): Control group: usual WIC care
  Interventions: Other: lifestyle intervention

INTERVENTIONS:
Other: lifestyle intervention

SUMMARY:
1) to evaluate treatment fidelity of DRRP: study design, training of interventionists, delivery and receipt of the intervention, and application of the intervention in real-life settings; 2) to identify successful strategies for participant recruitment and maintaining active participation; 3) to collect and analyze preliminary indicators of DRRP's effect on dietary intake, physical activity, stress responses, and body weight; and 4) To evaluate sample representativeness of the target audience, implementation and acceptability of DRRP, and attrition rate.

ELIGIBILITY:
Inclusion Criteria:Non-pregnant women between 18 and 34 years old who understood and spoke English and had a measured BMI between 25.0 and 39.9 kg/m2 were eligible for this study. Additional inclusion criteria included having a youngest child between 6 weeks and 3.5 years of age enrolled in one of our three collaborating WIC locations, not planning to become pregnant or change WIC clinics during the study, providing accurate contact information, agreeing to notify researchers with changes in contact information or pregnancy status, willingness to accept randomized participation assignments, being willing to participate in the project for 1.5 years, and consenting to have blood glucose tested via finger stick.

Exclusion Criteria: women with fasting blood glucose greater than 126 mg/dl or random blood glucose greater than 200 mg/dl, self-reported type 1 or 2 diabetes or an eating disorder, or inability to walk more than one block without resting or shortness of breath were excluded. Eligible participants provided their individual telephone and address and a telephone number of one back-up contact (relative, friend, or neighbor).

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult

PRIMARY OUTCOMES:
body weight

SECONDARY OUTCOMES:
dietary fat intake, fruit and vegetable intake, physical activity, stress, affects

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Michigan Stat University College of Nursing, East Lansing, Michigan
  - Michigan State University College of Nursing, East Lansing, Michigan

REFERENCES:
- [Derived] Chang MW, Brown R, Nitzke S. Participant recruitment and retention in a pilot program to prevent weight gain in low-income overweight and obese mothers. BMC Public Health. 2009 Nov 21;9:424. doi: 10.1186/1471-2458-9-424. PMID 19930587